CLINICAL TRIAL: NCT06256874
Title: Effect of Myofascial Release on Dysphagia Prevention for Elderly People in the Community: A Preliminary Self-control Study
Brief Title: Effect of Myofascial Release on Dysphagia Prevention for Elderly People in the Community
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Jinmo-old
Record Dates: First submitted 2024-02-03; First posted 2024-02-13 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the observation group (Experimental): The observation group is the only group of the participants.The elderly individuals will be arranged to undergo a continuous three-week (21 days) duration of Myofascial Release Training, with weekends off and training conducted only on weekdays, two sessions per day, each lasting 15-30 minutes. Each training session will be conducted approximately one hour prior to meals. Apart from this,we require participants to only engage in daily activities and avoid strenuous and dangerous behaviors
  Interventions: Behavioral: Myofascial Release Training

INTERVENTIONS:
Behavioral: Myofascial Release Training — Myofascial release, also known as fascial release or fascial manipulation, is a physical therapy used to treat muscle and fascial tissue tension or pain. It involves applying appropriate pressure and stretching to release tight fascia and soft tissues, improving blood circulation, alleviating pain, and promoting rehabilitation. Myofascial release therapy is commonly used to treat muscle spasms, chronic pain, skeletal and joint issues, among others.

SUMMARY:
The goal of this clinical trial is to explore the impact of Myofascial Release Training on swallowing function and quality of life in community-dwelling elderly individuals (≥60 year old) with swallowing disorders. It primarily aims to address the effects of Myofascial Release Training on swallowing function and quality of life in community-dwelling elderly individuals with swallowing disorders. All participants are required to undergo a continuous three-week (21 days) Myofascial Release Training, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 15-30 minutes each.

DETAILED DESCRIPTION:
Myofascial release, also known as fascial release or fascial manipulation, is a physical therapy used to treat muscle and fascial tissue tension or pain. It involves applying appropriate pressure and stretching to release tight fascia and soft tissues, improving blood circulation, alleviating pain, and promoting rehabilitation.

The goal of this clinical trial is to explore the impact of Myofascial Release Training on swallowing function and quality of life in community-dwelling elderly individuals (≥60 year old) with swallowing disorders. It primarily aims to address the effects of Myofascial Release Training on swallowing function and quality of life in community-dwelling elderly individuals with swallowing disorders. All participants are required to undergo a continuous three-week (21 days) Myofascial Release Training, with weekends off and training conducted only on weekdays. The training will be conducted two sessions per day, lasting 15-30 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years old.
* No hospitalization within the past six months.
* With clear consciousness and able to cooperate with questionnaires and training.
* The elderly people who voluntarily participate and agree to adhere until the end of the study.
* Dysphagia

Exclusion Criteria:

* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Physical disability.
* Difficulty in mobility.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Swallowing-Related Quality of Life Questionnaire | day 1 and day 21
  The Swallowing-Related Quality of Life Questionnaire (SWAL-QOL) is a validated tool used to assess the impact of swallowing difficulties on quality of life. It is a 44-item questionnaire designed to measure the physical, emotional, and social domains of swallowing-related quality of life.The higher final scores indicate the better life quality. The total score will be converted into a standard percentage

SECONDARY OUTCOMES:
Water Swallow Test | day 1 and day 21
  The Water Swallow Test was recruited to assess swallowing function in patients at admission. Specifically, patients were instructed to sit and drink 30 ml of warm water. A 5-point scoring system is used as follows:
  1. Point: Successful swallowing of water within 5 seconds without coughing.
  2. Points: Able to swallow the water once but taking more than 5 seconds or swallowing in two or more attempts without coughing.
  3. Points: Able to swallow the water once with coughing.
  4. Points: Able to swallow the water in two or more attempts with coughing.
  5. Points: Unable to swallow all of the water, frequent coughing. The higher points indicate the worse swallowing function
Time consumed in eating | day 1 and day 21
  We require participants to eat a lunch according to their daily intake and habits, and count the time consumed
Functional Oral Intake Scale | day 1 and day 21
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The Functional Oral Intake Scale assessment form includes seven levels of scoring, ranging from level 1 to level 7, indicating a progressive improvement in the patient's oral intake ability. In general, the result below level 6 indicates unsafe for oral intake while level 6 and above indicates that eating via mouth can be safely conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Chair — Site Coordinator of United Medical Group located in Miami
Locations (2):
- Taiwan (2):
  - Gaoxiong Rehabilitation Hospital, Xinzhu
  - Hsinchu Rehabilitation Hospital, Xinzhu

IPD SHARING:
Plan to Share IPD: No